CLINICAL TRIAL: NCT07021456
Title: Impact of Dietary Knowledge Related to Functional Insulin Therapy in Type 1 Diabetes on the Risk of Eating Disorders
Acronym: DIABEA
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Laboratoire TIMC-IMAG (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC24.0367; 2024-A02313-44 (Other: IDRCB)
Record Dates: First submitted 2025-02-24; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-04

CONDITIONS: Type 1 Diabetes (T1D)
Keywords: eating disorders; functional insulin therapy; type 1 diabetes; dietary knowledge
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Feeding and Eating Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Background: The management of type 1 diabetes (T1D) relies on exogenous insulin administration to compensate for the lack of endogenous insulin production. Optimal glycemic control, essential for preventing long-term complications, requires precise insulin dose adjustments based on carbohydrate intake. Functional insulin therapy (FIT) allows for flexibility in insulin dosing according to carbohydrate consumption, thereby reducing the dietary constraints previously imposed on patients. However, this approach requires increased attention to dietary intake. Individuals with T1D already have a heightened risk of developing eating disorders (EDs). We hypothesize that the dietary knowledge required for FIT may contribute to rigid eating behaviors, thereby increasing the risk of EDs.

Objective: This prospective monocentric study aims to determine whether dietary knowledge related to FIT is associated with an increased risk of EDs in individuals with T1D.

Methods: The primary outcome measure is the correlation between the Gluciquizz score (a validated tool assessing FIT knowledge) and the risk of EDs, evaluated using the DEPS-R questionnaire (a validated screening tool for ED risk in T1D patients). In addition to this quantitative analysis, a qualitative study will be conducted through semi-structured interviews to explore in greater depth the patients' experiences, their relationship with food, and their perceptions of FIT-related requirements.

Perspectives: This study aims to improve the understanding of the impact of FIT on ED risk in T1D. The findings may help identify at-risk patient profiles and enhance therapeutic education and patient management by integrating ED risk considerations. The qualitative approach will provide further insight into patients' individual experiences, facilitating recommendations tailored to their specific needs.

DETAILED DESCRIPTION:
STUDY DESCRIPTION

This is a Type 3 study under the Jardé law, involving human subjects:

Observational study Prospective design Monocentric National scope

We selected this study design to minimize participant burden (data collection conducted online, by phone, or via videoconference, eliminating the need for patient travel). Recruitment through patient association websites and social media will enable a national reach.

The study will take place in four phases:

Recruitment Videoconference for a questionnaire on FIT-related dietary knowledge and ED risk assessment Self-administered online questionnaire Videoconference interview

SELECTION AND INCLUSION VISIT

If the participant wishes to join the study, they can either scan the QR code or visit the web link provided in the recruitment announcement. This QR code or link will redirect to a page detailing the study, the eligibility criteria that the participant must complete, and the information notice. The participant will enter their email address in the designated field and will also have the option to download the information notice if they wish.

Once this step is completed, the principal investigator will verify the eligibility criteria. If the participant meets the criteria, they will receive an email containing the necessary information for the next steps of the study:

Non-opposition letter - Part 1 A personal identifier number (formatted as initials + number, e.g., LA01) to pseudonymize questionnaire and self-reported responses A calendar allowing them to indicate their preferred date for the videoconference A link to access the videoconference

To ensure that the participant fully understands the study procedures, the clinical research associate (CRA) will go over the project details during the first videoconference and address any questions. The CRA will also check that the non-opposition form has been properly completed before integrating it into the study records.

If the participant does not meet the eligibility criteria, they will receive an email notifying them of their ineligibility.

The principal investigator will maintain a correspondence table containing the participant's name, surname, email address, and personal identifier number.

Participants will be fully and transparently informed in clear and understandable terms about the study objectives, the nature of the collected data, and their right to withdraw their consent at any time. The investigator must also inform participants about the opinion issued by the Ethics Committee (Comité de Protection des Personnes - CPP).

Participants can exercise their right to oppose the processing of their health data for research purposes at any time by contacting either the research coordinator or the institution responsible for the data. The institution is committed to responding to such requests within a maximum of two months.

FOLLOW-UP VISITS

The study will be conducted in three distinct phases:

1. First Phase: Videoconference for Questionnaire Completion

   A clinical research associate (CRA) will contact the participant to administer the questionnaires. The CRA will directly enter the participant's responses into the Redcap online platform.

   At the end of this interview, the investigator will invite participants to take part in the qualitative phase of the study (third phase: semi-structured videoconference interview). Participants will be progressively included until data saturation is reached.

   If the participant agrees, the investigator will send a second email with a second non-opposition form - Part 2 (Appendix 4) for participation in the qualitative interview.

   For all participants, a Redcap platform link will be emailed to them to complete the self-reported questionnaires.
2. Second Phase: Online Self-Questionnaires

   Participants will receive a link to complete self-administered questionnaires directly on Redcap. Contact information for the CRA or investigator will be provided in case of technical issues.
3. Third Phase: Semi-Structured Videoconference Interview

This interview will be semi-structured and will follow the interview guide provided in Appendix 12. Participants will be included in this phase until data saturation is reached.

For the first and third phases, we have chosen to conduct interviews via the BigBlueButton videoconferencing platform, which is GDPR-compliant. We aim to use a platform that is user-friendly and free for participants.

Since BigBlueButton is integrated with the Université Grenoble Alpes information system, no additional identification data will be processed. The following personal data-voice and image-will be recorded by the interview organizer.

If the recording feature is activated, participants will be explicitly notified via a specific message. The recordings will be used exclusively for the transcription of data.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 1 diabetes confirmed by a referring physician
* Diagnosis received at least three months prior
* Adult (18 years or older)
* Access to a computer or smartphone capable of videoconferencing
* No expressed opposition to participation
* Consent for image rights (for Phase 2 qualitative interviews)

Exclusion Criteria:

* Inability to complete online questionnaires and participate in a 45-minute videoconference interview
* Being under legal guardianship or curatorship
* Being pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We aim to include patients with type 1 diabetes (T1D) in France. Participants will be enrolled in the study regardless of their current treatment.
  We will reach out to French patient associations for individuals with T1D, such as the Fédération Française des Diabétiques, to request the dissemination of our recruitment announcement to their members. The announcement will also be published on social media. Recruitment will be based on an online announcement, attached in Appendix 1.
  Additionally, we will propose to the Endocrinology Department at CHU Grenoble-Alpes to display the recruitment announcement in their waiting rooms to present it to their patients. If these recruitment channels do not yield a sufficient number of participants, we will expand dissemination to other hospital departments at the national level.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
to determine whether dietary knowledge related to functional insulin therapy (FIT) is associated with the risk of developing eating disorders (EDs) | Day 1
  the correlation between the Gluciquizz score (a validated tool assessing FIT knowledge) and the risk of EDs, as measured by the DEPS-R questionnaire.

SECONDARY OUTCOMES:
To determine whether dietary knowledge related to FIT is associated with the risk of EDs according to the SCOFF-F questionnaire (a validated French screening tool for EDs). | Day 1
  Correlation between the Gluciquizz score (validated for assessing FIT knowledge) and the risk of EDs according to the SCOFF-F questionnaire.
To assess whether the following factors influence the risk of developing EDs: a. Quality of life | Day 1
  Comparison of the following factors: quality of life (measured by ADDQoL, unit: individual weighted impact score) between two groups defined by the DEPS-R threshold (≤ 20 vs. > 20, indicating ED risk).
To identify whether specific patient profiles at risk of developing EDs emerge based on the collected variables. | Day 1
  Identification of patient profiles based on the following variables: FIT knowledge (Gluciquizz, unit: percentage of correct responses), quality of life (ADDQoL, unit: individual weighted impact score), diabetes-related anxiety (PAID, unit: total score ranging from 0 to 100), fear of hypoglycemia (HFS-II, unit: total score ranging from 0 to 33 for the behavior subscale and 0 to 45 for the worry subscale), diabetes duration (unit: years), and treatment (unit: type of treatment, e.g., insulin therapy, oral antidiabetic drugs), with DEPS-R (unit: total score ranging from 0 to 30) as an illustrative variable.
To explore the influence of functional insulin therapy on eating behaviors through semi-structured interviews. | Day 1
  Insights into the decision-making factors influencing food choices among individuals with type 1 diabetes, following qualitative study methodologies.
To assess whether the following factors influence the risk of developing EDs: b. Diabetes-related anxiety | Day 1
  Comparison of the following factors: diabetes-related anxiety (PAID, unit: total score ranging from 0 to 100) between two groups defined by the DEPS-R threshold (≤ 20 vs. > 20, indicating ED risk).
To assess whether the following factors influence the risk of developing EDs: c. fear of hypoglycemia | Day 1
  Comparison of the following factors: fear of hypoglycemia (HFS, unit: total score ranging from 0 to 8) between two groups defined by the DEPS-R threshold (≤ 20 vs. > 20, indicating ED risk).

CONTACTS AND LOCATIONS:
Locations (1):
- Grenoble, Grenoble, France

REFERENCES:
- [Background] De Paoli T, Rogers PJ. Disordered eating and insulin restriction in type 1 diabetes: A systematic review and testable model. Eat Disord. 2018 Jul-Aug;26(4):343-360. doi: 10.1080/10640266.2017.1405651. Epub 2017 Nov 28. PMID 29182474
- [Background] Palmieri S, Mansueto G, Ruggiero GM, Caselli G, Sassaroli S, Spada MM. Metacognitive beliefs across eating disorders and eating behaviours: A systematic review. Clin Psychol Psychother. 2021 Sep;28(5):1254-1265. doi: 10.1002/cpp.2573. Epub 2021 Feb 23. PMID 33606916
- [Background] Cheng R, Taleb N, Stainforth-Dubois M, Rabasa-Lhoret R. The promising future of insulin therapy in diabetes mellitus. Am J Physiol Endocrinol Metab. 2021 May 1;320(5):E886-E890. doi: 10.1152/ajpendo.00608.2020. Epub 2021 Mar 15. PMID 33719586